CLINICAL TRIAL: NCT03268148
Title: Analgesic Effect of Low Level Laser for Procedural Pain in Newborn Infants: an Open-label, Randomized-controlled Trial
Brief Title: Analgesic Effect of Low Level Laser for Procedural Pain in Newborn Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Bei-yu Wu, Atteding doctor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201700474A3C501
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Procedural Pain
Keywords: neonates; pain; low level laser
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: low level laser group and breast milk group
Who Masked: Outcomes Assessor
Masking Description: Two independent assessors blinded to intervention read the video, and then record vital signs and pain score. The videos are cut from heel-lancing to the end so that the assessors do not know whether the neonate receive low level laser or breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low level laser group (Experimental): LaserPen is applied to the local point for 20 seconds where heel-lancing will be performed in the low level laser group.
  Interventions: Device: LaserPen
- breast milk group (No Intervention): Subjects in breast milk group are given 5ml expressed breast milk by mouth using a syringe tube inserted to the participant's oral cavity over a 2-minute period before heel-lancing.

INTERVENTIONS:
Device: LaserPen — low level laser is used before heel-lancing for newborn screening
  Other Names: power 150mW, wavelength 810nm, RJ-laser
  Arms: low level laser group

SUMMARY:
Neonates undergo several painful procedures and these pain experiences can alter clinical outcome and behavior. The investigators aim to investigate the analgesic effect of low level laser for procedural pain during heel lancing of term neonates.

DETAILED DESCRIPTION:
This open-label, randomized controlled trial involves 130 term newborn infants (gestational ages between 37 weeks to 42 weeks) who need heel lancing for newborn screening. Subjects are randomly assigned to low level laser group or breast milk group. Subjects in breast milk group are given 5ml expressed breast milk by mouth using a syringe tube inserted to the participant's oral cavity over a 2-minute period. LaserPen is applied to the local point for 20 seconds where heel-lancing will be performed in the low level laser group. Then heel lancing is performed and two observers who are blinded to the intervention record the physiological (heart rate and oxygen saturation) and behavioral parameters (duration of crying and modified neonatal facial coding scores) following the procedure. Heart rate variation of participants is record by CheckMyHeart ECG monitor. The salivary swab method is used to detect the infant's salivary cortisol and amylase level as biomarker for stress evaluation. During the study course, digital cameras continuously record participants' behavior. Independent t-test, chi-squared test and one way ANOVA are used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* healthy fullterm neonates (37-42 gestational age)
* Apgar score >= 7
* will receive newborn screening

Exclusion Criteria:

* >42 or < 37 gestational age
* perinatal asphyxia
* major malformations or any other disease that need intensive care
* drug withdrawal received previous treatment

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
pain assessment | immediately after heel-lancing
  latency of first cry, crying time, squeezing time, neonatal facial coding system(NFCS), Neonatal Pain, Agitation and Sedation Scale (NPASS)

SECONDARY OUTCOMES:
stress biomarker | baseline, immediately after heel-lancing, 20 minutes after heel-lancing
  The salivary swab method is used to detect the infant's salivary cortisol and amylase level at 3 time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bei-yu Wu, doctor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ou-Yang MC, Chen IL, Chen CC, Chung MY, Chen FS, Huang HC. Expressed breast milk for procedural pain in preterm neonates: a randomized, double-blind, placebo-controlled trial. Acta Paediatr. 2013 Jan;102(1):15-21. doi: 10.1111/apa.12045. Epub 2012 Nov 1. PMID 23057434